CLINICAL TRIAL: NCT01043835
Title: Prospective Randomized Trial of Laparoscopic Versus Open Gastrectomy for Advanced Gastric Cancer
Brief Title: Comparison of Laparoscopic Versus Open Gastrectomy for Advanced Gastric Cancer:A Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yan Shi (Other)
Responsible Party: Sponsor-Investigator, Yan Shi, Department of General Surgery and Center of Microinvasive Gastrointestinal Surgery, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197691197392
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Stomach Neoplasm; Laparoscopy; Gastrectomy; Complications
Keywords: Stomach Neoplasm; Laparoscopy; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopy-assisted gastrectomy (Experimental)
  Interventions: Procedure: Laparoscopy-assisted gastrectomy
- Open gastrectomy (Active Comparator)
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopy-assisted gastrectomy — A 10-mm trocar for laparoscope was inserted below the umbilicus. Another 10-mm trocar was introduced in the left preaxillary line 2 cm below the costal margin as a major hand port，and a 5-mm trocar was placed at the contralateral site for traction. A 5-mm trocar was inserted in the left midclavicular line 2 cm above the umbilicus as an accessory port, and a 15-mm trocar also as an accessory port was placed at the contralateral site. The operator stood on the left side of the patient. Subtotal or total gastrectomy and D2 lymph node dissection will be performed basically. As a general rule, Billroth I, Billroth II or Roux-Y method was used for gastric reconstruction. Dissected stomach and lymph node are collected through additional 5 cm incision at a median superior abdominal incision.
  Arms: Laparoscopy-assisted gastrectomy
Procedure: Open gastrectomy — Approximately 15~20 cm length incision is made from falciform process to periumbilical area. Subtotal or total gastrectomy and D2 lymph node dissection will be performed basically. As a general rule, Billroth I, Billroth II or Roux-Y method was used for gastric reconstruction for all cases.
  Arms: Open gastrectomy

SUMMARY:
The purpose of this study is to compare the short- and long-term results between the laparoscopy-assisted gastrectomy and the open gastrectomy.

DETAILED DESCRIPTION:
Background: The use of laparoscopic surgery in the management of advanced gastric cancer (AGC) has not yet met with widespread acceptance and remains limited to only a few centers.

Intervention: According to tumor pathological stage (JGCA, 2nd English ed), location of tumor, and patient clinical condition, a laparoscopy-assisted radical gastrectomy and open gastrectomy were performed. Laparoscopy-assisted radical gastrectomy consisted of the following procedures: 1) laparoscopic dissection of the lesser and greater omentum, ligation and division of the main vessels to mobilize the stomach under pneumoperitoneum, 2) laparoscopic D2 lymph node dissection, based on the Guidelines of the Japan Gastric Cancer Association and 3) resection of the distal two thirds (LADG), proximal third (LAPG), or total stomach (LATG), depending on the location of the tumor, followed by reconstruction by the Billroth I, Billroth Ⅱ, esophagogastrostomy, or Roux-en-Y method through a 3 to 5-cm-long minilaparotomy incision.

Follow-up schedule: All patients were monitored postoperatively by physical examination, and blood tests including a test for serum carcinoembryonic antigen (CEA) at least every three months for the ﬁrst year, every six months for the next two years, and every year for the fourth and fifth year, and thereafter by abdominal ultrasonography, CT, chest radiography, and gastroscopy at least once each year.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven gastric adenocarcinoma
2. Age:older than 18 years old,younger than 80 years old
3. Preoperative stage(CT, GFS stage):cT2N0M0, cT2N1M0, cT2N2M0, cT3N0M0, cT3N1M0,cT3N2M0
4. ASA score:≤3
5. Patients with an invasion of the gastric serosa exceeding 10 cm2 according to ultrasound examination or examination during surgery were excluded
6. No history of other cancer
7. No history of chemotherapy or radiotherapy
8. Written informed consent

Exclusion Criteria:

1. Concurrent cancer patients or patient who was treated due to other types of cancer before the patient was diagnosed as a gastric cancer patient
2. Patient who was treated by other types of treatment methods, such as chemotherapy, immunotherapy, or radiotherapy
3. Patient who was received upper abdominal surgery (except, laparoscopic cholecystectomy)
4. ASA score:>3
5. Contraindication of laparoscopy: severe cardiac disease, abdominal wall hernias, diaphragmatic hernias, uncorrected coagulopathies, portal hypertension, pregnancy
6. Complicated case needed to get emergency operation
7. Any accompanying surgical condition needed to be performed in same time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2010-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years

SECONDARY OUTCOMES:
Complications, recurrence, quality of life measured by EORTC QLQ-C30 V 3.0 and EORTC QLQ-STO22 | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of General Surgery and Center of Microinvasive Gastrointestinal Surgery, Southwest Hospital, Chongqing, Chong Qing
  - Southwest Hospital, China, Chongqing, Chong Qing